CLINICAL TRIAL: NCT06204731
Title: The Influence of Physical Training in Normobaric Hypoxia on Prooxidant-Antioxidant Imbalance, Inflammatory Marker Levels, Intestinal Damage Degree, and Mitochondrial Energy Release Rate in Young Non-trained Males
Brief Title: The Impact of Physical Training Under Normobaric Hypoxia on Oxidative Stress Level, Inflammatory State, Intestinal Damage, and Mitochondrial Metabolism in Young Males
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University School of Physical Education, Krakow, Poland (Other)
Collaborators: Ministry of Education and Science,Poland (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SKN/SP/570048/2023
Record Dates: First submitted 2023-12-11; First posted 2024-01-12 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2023-12

CONDITIONS: Hypoxia, Altitude
Keywords: inflammation; oxidative stress; intestinal damage; muscle damage; mitochondrial metabolism; normobaric hypoxia; training
MeSH Terms: conditions — Altitude Sickness; Inflammation | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group (No Intervention): The control group will not undergo the training program.
- LHTL (live high - train low) (Experimental): Training performed under normoxic conditions (223m), stay and sleep in normobaric hypoxic conditions (3000m) and thermoneutral conditions (21°C) and constant humidity (40%).
  Interventions: Other: Exercise and environmental conditions
- LLTH (live low - train high) (Experimental): Training performed under normobaric hypoxia conditions (3000m), stay and sleep in normoxic conditions (223m) and thermoneutral conditions (21°C) and constant humidity (40%).
  will stay and sleep in normoxic (223m), and train in normobaric hypoxia (3000m)
  Interventions: Other: Exercise and environmental conditions
- LLTL (live low - train low) (Experimental): Training performed and stay and sleep in normoxic conditions (223m) and thermoneutral conditions (21°C) and constant humidity (40%).
  Interventions: Other: Exercise and environmental conditions

INTERVENTIONS:
Other: Exercise and environmental conditions — Participants will engage in interval training and will reside and sleep at different altitudes for a period of 4 weeks. Aerobic and anaerobic capacity tests and an eccentric exercise test will be performed before and after the training intervention. Before and after the training program, somatic measurements will also be taken. Before and after the first and last workout, blood will be drawn for biochemical analysis.
  Arms: LHTL (live high - train low); LLTH (live low - train high); LLTL (live low - train low)

SUMMARY:
* Cognitive assessment of the influence of a 4-week proprietary training program under normobaric hypoxia conditions on the levels of inflammatory markers, disturbances in prooxidant-antioxidant balance, degree of intestinal damage, and mitochondrial energy production rate in young sedentary males.
* Applied objective: Development of practical training guidelines utilizing training in normobaric hypoxia conditions to enhance mechanisms related to oxygen transport, adaptive changes within the immune system, body's antioxidant capacity, gut permeability, substrate utilization efficiency, and mitochondrial function for coaches and athletes.

ELIGIBILITY:
Inclusion Criteria:

* no known metabolic diseases, no contraindications to physical exercise and no history of high altitude sickness stated in interview. A medical examination (including ECG, blood and urine tests) is required.

Exclusion Criteria:

* changes in diet during the experiment, smoking and abuse of alcohol and/or other stimulants.

Ages: 19 Years to 29 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Measurement of aerobic capacity (endurance) | 7 days before training and 7-10 days after the training. Training will last 4 weeks.
  Measurement of maximal oxygen uptake and determination of ventilatory thresholds (ergospirometry)
Measurement of anaerobic capacity | 7 days before training and 7-10 days after the training. Training will last 4 weeks
  Measurement of maximal anaerobic power (Wingate Anaerobic Test)
Blood analysis | 7 days before training and 7- 10 days after the training. The training will last 4 weeks and will consist of 12 workouts.
  Indicators of prooxidant-antioxidant imbalance, markers of inflammatory status, markers of muscle damage, markers of intestinal damage, HIF (hypoxia-inducible factor), EPO (erythropoietin), markers of mitochondrial metabolism, morphology (including reticulocytes).
Somatic indices | 7 days before training and 7-10 days after the training. Training will last 4 weeks.
  Body composition analysis ( body height [m], body mass [kg], Quetelet II Index [kg/m^2], lean body mass [kg], fat mass [kg], fat percentage [%] and total water content [kg]

CONTACTS AND LOCATIONS:
Locations (1):
- University School of Physical Education in Cracow, Krakow, Poland

IPD SHARING:
Plan to Share IPD: No